CLINICAL TRIAL: NCT01183247
Title: An Open, Single Centre, Randomised, Parallel Group Study to Investigate Three Different Immunosuppressive Regimens for de Novo Renal Transplant Recipients: A Comparison of a Sirolimus / EC-MPS (Myfortic) / Tacrolimus Regimen, an Everolimus / EC-MPS / Tacrolimus Regimen and a EC-MPS / Tacrolimus Prednisone Regimen
Brief Title: An Open, Single Centre, Randomised, Parallel Group Study to Investigate Three Different Immunosuppressive Regimens
Acronym: SterFreePlus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Novartis (Industry)
Responsible Party: Juerg Steiger, professor, clinic for transplantation immunology and nephrology, university hospital Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187/07
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Comparative Study; Immunosuppressive Agents
Keywords: Everolimus,; rapamycin,; prednisone,; tacrolimus,; MMF,; steroid-free,; protocol biopsy
MeSH Terms: interventions — Sirolimus; Everolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rapamycin (Active Comparator): Rapamycin-MMF-tacrolimus
  Interventions: Drug: Rapamycin
- Everolimus (Active Comparator): Everolimus - tacrolimus - MMF
  Interventions: Drug: Everolimus
- Prednisone (Active Comparator): tacrolimus - MMF -prednisone
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Rapamycin — Add rapamycin de novo to tacrolimus and MMF
  Other Names: Sirolimus
  Arms: Rapamycin
Drug: Everolimus — Add everolimus de novo to tacrolimus and MMF
  Arms: Everolimus
Drug: Prednisone — Add prednisone de novo to tacrolimus and MMF
  Arms: Prednisone

SUMMARY:
An open, single center, randomised study to investigate three different immunosuppressive regimens for de novo renal transplant recipients:

1. st sirolimus / EC-MPS / tacrolimus regimen

   - After 3 months a protocol biopsy is performed. If no rejection is detected the calcineurin inhibitor (tacrolimus) is withdrawn.
2. nd everolimus / EC-MPS / tacrolimus regimen

   - After 3 months a protocol biopsy is performed. If no rejection is detected the calcineurin inhibitor (tacrolimus) is withdrawn.
3. rd tacrolimus / EC-MPS / prednisone regimen - After 3 months a protocol biopsy is performed. If no rejection is detected prednisone is withdrawn.

DETAILED DESCRIPTION:
This study is designed to show similar efficacy but a different adverse event profile between the three regimens. Its main purpose is to provide more information, if steroid free immunosuppressive treatment is a valuable alternative in the treatment of de novo kidney transplant recipients and that it is possible to withdraw calcineurin inhibitors after 3 months in this steroid free protocol. A secondary rationale of the study is to compare sirolimus with everolimus directly to better differentiate these two mTOR-inhibitors in terms of compound-specific effects and class-effects. This should allow for early conclusions on the usage of these two mTOR-inhibitors in CNI-free regimens.

Basis for this study are the following hypotheses regarding the first 6 months of treatment following kidney transplantation:

* Similar graft function in the three treatment groups after 6 months
* No difference in graft and patient survival in the three groups
* No differences in incidence of first, total number, type of acute rejections, and number of anti-rejection treatments in the three groups
* No differences in number of patients successfully withdrawn from calcineurin inhibitor in the sirolimus and everolimus arm, respectively
* A different adverse event profile with regard to the incidence of dyslipidemias, impaired fasting glucose, new onset diabetes mellitus, de novo post-transplant insulin dependency, histological signs of calcineurin inhibitor toxicity, and tubulointerstitial nephrotoxicity in the three groups. In addition to this the incidence of mTOR-inhibitor specific adverse events will be analysed.

These hypotheses are the basis for the study objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 75 years of age, regardless of race.
2. Female patients of child bearing age agree to maintain effective birth control practice during the study.
3. Patient has end stage kidney disease and is a suitable candidate for primary renal transplantation or retransplantation as assessed by the transplantation centre.
4. Patient has been fully informed and has given written or independent person witnessed oral informed consent.

Exclusion Criteria:

1. in Patient is pregnant or breastfeeding.
2. Patient has a low immunological risk constellation, defined by receiving a kidney from a HLA-identical related living donor.
3. Patient has a high immunological risk constellation, defined as having donor specific HLA-antibodies and/or having a previous graft survival shorter than 3 years due to rejection.
4. Patient and donor have a positive T or B-cell crossmatch.
5. Patient and donor are ABO incompatible.
6. Age of donor > 75 years.
7. Cold ischemia time > 36 hours.
8. Patient has leucopenia, defined as having at transplantation less than 3000/mm3 leukocytes.
9. Patient has thrombocytopenia, defined as having at transplantation less than 75000/mm3 thrombocytes.
10. Patient is allergic or intolerant to cremophor RH 60 or structurally related compounds, steroids, everolimus, tacrolimus, Sirolimus or EC-MPS.
11. Patient or donor is known to be HIV positive.
12. Patient has significant liver disease, defined as having during the past 28 days continuously ASAT (SGOT) and/or ALAT (SGPT) levels greater than 3 fold of the upper value of the normal range of the investigational site.
13. Patient with malignancy or history of malignancy ≤ 2 years, except non metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
14. Patient has significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, or active peptic ulcer.
15. Patient is taking or has been taking an investigational drug in the past 28 days.
16. Patient has previously received or is receiving another organ transplant other than kidney.
17. Patient is unlikely to comply with the visits schedule the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Plasma creatinine and creatinine clearance (Cockcroft-Gault) after 6 months of treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Juerg U Steiger, Professor, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinic for transplantation immunology and nephrology, Basel, Switzerland